CLINICAL TRIAL: NCT06185335
Title: An Open-Label Two-Stage Trial of the Safety, Pharmacodynamics, Biodistribution, Immunogenicity and Efficacy of Single-Dose Administration of ANB-010 in Subjects With Hemophilia A
Brief Title: A Trial of the Safety and Efficacy of Single-Dose Administration of ANB-010 in Subjects With Hemophilia A
Acronym: EDELWEISS
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ANB-010-1
Record Dates: First submitted 2023-12-01; First posted 2023-12-29 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1 (Experimental): Subjects in Cohort 1 will receive ANB-010 at a dose 1. ANB-010 will be administered to the first subject in group 1. Not earlier than in 28 days, the investigational product will be administered to the next two subjects in Cohort 1 (with an interval of at least 24 hours).
  Interventions: Genetic: ANB-010, dose 1
- Cohort 2 (Experimental): Subjects in Cohort 2 will receive ANB-010 at a dose 2. Not earlier than 28 days after the ANB-010 administration to the third subject in Cohort 1, the investigational product will be administered to the first subject in Cohort 2. Not earlier than 28 days after the ANB-010 administration to the first subject in Cohort 2, the investigational product will be administered to the next two subjects in Cohort 2 (with an interval of at least 24 hours).
  Interventions: Genetic: ANB-010, dose 2
- Cohort 3 (Experimental): Subjects in Cohort 3 will receive ANB-010 at a dose 3. Not earlier than 28 days after the ANB-010 administration to the third subject in Cohort 2, the investigational product will be administered to the first subject in Cohort 3. Not earlier than 28 days after the ANB-010 administration to the first subject in Cohort 3, the investigational product will be administered to the next two subjects in Cohort 3 (with an interval of at least 24 hours).
  Interventions: Genetic: ANB-010, dose 3

INTERVENTIONS:
Genetic: ANB-010, dose 1 — Adeno-associated viral vector carrying the FVIII gene single infusion at dose 1.
  Arms: Cohort 1
Genetic: ANB-010, dose 2 — Adeno-associated viral vector carrying the FVIII gene single infusion at dose 2.
  Arms: Cohort 2
Genetic: ANB-010, dose 3 — Adeno-associated viral vector carrying the FVIII gene single infusion at dose 3.
  Arms: Cohort 3

SUMMARY:
The goal of this multicenter, two-stage, open-label study is to investigate the safety, immunogenicity, and efficacy of ANB-010 in subjects with hemophilia A. The study will have a dose-escalation design with elements of phase I/II seamless adaptive design.

DETAILED DESCRIPTION:
The study will be conducted in 2 stages:

Stage 1: pilot efficacy and safety study of different doses to select a potentially therapeutic dose for further study.

Stage 2: study of the efficacy and safety of ANB-010 at the selected potentially therapeutic dose.

The stage 1 design is typical of phase I clinical trials with a modified "3+3" design and dose escalation. Three subjects are to be sequentially included in each cohort, each of whom will recieved a pre-specified cohort dose of ANB-010 as a single inravenous infusion.

Subjects will be monitored for dose-limiting toxicity (DLT) events for 4 weeks after the drug infusion. The decision concerning dose escalation will be made at the Independent Data Monitoring Committee (IDMC) meetings.

At the second stage the main study period will include 6 subjects who will receive ANB-010 at the optimal dose selected based on the results of stage 1 data analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects aged ≥18 years at the time of signing the informed consent form.

3. Established diagnosis of hemophilia A with a documented history of endogenous FVIII activity ≤1% AND ≤2% at screening.

4. Therapy with FVIII concentrates for at least 150 exposure days.

Exclusion Criteria:

1. History of use of any gene therapy product.
2. Use of emicizumab within less than 6 months before the date of signing the ICF.
3. The presence of other blood or hematopoietic disorders other than hemophilia A.
4. Presence of AAV6 antibodies detected by ELISA.
5. BMI <16 kg/m² or ≥35 kg/m².
6. Diagnosis of HIV infection.
7. HBV infection.
8. HCV infection.
9. Any active systemic infections or recurrent infections requiring systemic therapy at screening.
10. Any other disorders associated with severe immunodeficiency.
11. Relevant hepatic disorders or conditions that can be a symptom of existing liver disorder.
12. Malignancies with remission duration of less than 5 years at the time of signing the ICF, except for cured basal cell carcinoma.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-07-26 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2033-06 (Estimated)

PRIMARY OUTCOMES:
Change in FVIII activity from baseline to Week 52 | 12 months
Assessment of ANB-010 safety | 12 months
  Proportion and characteristics of adverse events

SECONDARY OUTCOMES:
Change in FVIII activity from baseline to scheduled assessment visits | 12 months
  FVIII activity will be assessed at every scheduled visits and compared to baseline
Proportion of subjects achieving clinical response | 12 months
  Clinical response is formulated as FVIII activity of 5-150%
Proportion of subjects who achieved normalized response | 12 months
  Normalized response is formulated as FVIII activity of 50-150%
Annualized consumption of FVIII concentrates by a subject | 12 months
Annualized bleeding rate | 12 months
Annualized rate of bleeding requiring therapy with FVIII concentrates | 12 months
Duration of response based on activity FVIII | 12 months

OTHER OUTCOMES:
Pharmacodynamics of ANB-010 | 12 months
  Evaluation of peak and steady-state FVIII concentrations
Proportion of subjects with FVIII inhibitor | 12 months
Proportion of subjects with antibodies to capsid | 12 months
Proportion of subjects with anti-FVIII antibodies | 12 months
Proportion of subjects with T cells specific to AAV6 and FVIII transgene product | 12 months
ANB-010 biodistribution (in blood, saliva, urine, semen and feces) | 12 months
Annualized rate of spontaneous bleeding | 12 months
Annualized rate of intraarticular bleeding | 12 months
Annualized rate of trauma-related bleeding | 12 months
Change from baseline in the quality of life measured with Haemo-A-QoL | 12 months
  The assessment will be provided at scheduled assessment visits (if the scale is available in the CS).
Change from baseline in the quality of life measured with EuroQol-5D-3L | 12 months
  The assessment will be provided at scheduled assessment visits (if the scale is available in the CS).
Change from baseline in the quality of life measured with SF-36 | 12 months
  The assessment will be provided at scheduled assessment visits (if the scale is available in the CS).
Change from baseline in the assessment on the Health Needs Questionnaire for Adults with Hemophilia A at scheduled assessment visits | 12 months
  The assessment is be performed if the scales are available in the CS.
Joint assessment based on HJHS v.2.1 | 12 months
  The assessment is be performed if the scales are available in the CS.

CONTACTS AND LOCATIONS:
Overall Officials: Arina V Zinkina-Orikhan, PhD, Study Director — Director of Clinical Development Department, BIOCAD
Locations (17):
- Russia (17):
  - State Autonomous Institution for Healthcare "Chelyabinsk Regional Clinical Hospital", Chelyabinsk
  - State budgetary healthcare institution Leningrad Regional Clinical Hospital, Gatchina
  - Kuzbass Clinical Hospital named after S.V. Belyaev, Kemerovo
  - Federal State Budgetary Organization of Science "Kirov Research Institute of Hematology and Blood Transfusions of Federal Medical Biological agency", Kirov
  - Federal State Budgetary Institution "National Medical Research Centre for Hematology" of the Ministry of Health of Russian Federation (Department of Clinical Diagnostics for Hematology and Hemostasis Disorders), Moscow
  - Federal State Budgetary Institution "National Medical Research Centre for Hematology" of the Ministry of Health of Russian Federation (Department of Traumatology and Reconstructive and Restorative Orthopedics for Patients with Hemophilia), Moscow
  - Research Center for Hematology MHSD RF, Moscow
  - Federal Budgetary Institution "Moscow City Clinical Hospital named after S. P. Botkin", Moscow
  - LLC "Medis", Nizhny Novgorod
  - State Novosibirsk Regional Clinical Hospital, Novosibirsk
  - Russian Research Institute of Hematology and Transfusiology Federal State Institution of Federal Medical and Biological Agency, Saint Petersburg
  - City Polyclinic №37, Saint Petersburg
  - Almazov National Medical Research Centre, Saint Petersburg
  - Federal State Budgetary Educational Institution of Higher Education "Samara State Medical University" of the Ministry of Healthcare of the Russian Federation, Samara
  - State Institution "Komi Republican Oncological Dispensary", Syktyvkar
  - Federal State Budgetary Educational Institution of Higher Education "Bashkir State Medical University" of the Ministry of Healthcare of the Russian Federation, Ufa
  - State Autonomous Institution for Healthcare of Sverdlovsk region "Sverdlovsk Regional Clinical Hospital №1", Yekaterinburg

IPD SHARING:
Plan to Share IPD: No